CLINICAL TRIAL: NCT03406390
Title: The Effects of Primary Pterygium on Contrast Sensitivity Preoperatively and Postoperatively
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2017011
Record Dates: First submitted 2017-11-03; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Primary Pterygium
Keywords: contrast sensitivity; Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primary pterygium: Observe the contrast sensitivity of primary pterygium patients and healthy control by quick CSF methods, and the pterygium group would achieve the pterygium surgery by the same surgeon (Jin Yuan) and then be performed the contrast sensitivity test on the 1st, 3rd and 6th month postoperatively.
  Interventions: Procedure: Pterygium surgery

INTERVENTIONS:
Procedure: Pterygium surgery — The patients were anesthetized with subconjunctival injection.Symblepharon was released and fibrotic tissue was extensively dissected to expose the sclera and corneal stroma. The subconjunctival fibrovascular tissue, including Tenon's capsule, were thoroughly removed using scissors from the sclera and medial rectus muscle at the area of the superior and inferior fornices and the nasal caruncle. A cryopreserved human amniotic membrane (Zhongshan Ophthalmic Center, China) was then placed on the entire exposed bare sclera with the epithelial side facing upward, and secured with 10-0 nylon sutures.

SUMMARY:
Pterygium is the growth of conjunctival tissue onto the cornea, usually from the nasal quadrant of the cornea.Visual acuity may be reduced due to direct invasion of the visual axis or astigmatism induced by the pterygium. Contrast sensitivity measures two variables, size, and contrast which could comprehensively reflect the visual quality of the primary pterygium patients. In this study, we would investigate the the effects of primary pterygium on contrast sensitivity preoperatively and on the 1st, 3rd and 6th month postoperatively, moreover, the related parameters on the contrast sensitivity in the primary pterygium patients would be analyzed.

DETAILED DESCRIPTION:
There would have two groups included in our study, which are primary pterygium group(40 patients) and the normal group (20 volunteers). The inclusion criteria for the primary pterygium group were: 1) more than 18 and less than 60 years old; 2)diagnosed as primary pterygium by the professional doctor; 3)0.0 or better logMAR BCVA; 4) absence of other ocular disorders and no history of eye surgery and other systemic diseases. The inclusion criteria for the normal group were: 1) between 18 and 60 years old; 2) 0.0 or better logMAR BCVA;3) no history of any ocular pathology, and normal physical and mental health.

All the subjects would receive the ophthalmic examination and contrast sensitivity test (quick contrast sensitivity function, quick CSF), in which the pterygium group would achieve the pterygium surgery by the same surgeon (Jin Yuan) and then be performed the contrast sensitivity test on the 1st, 3rd and 6th month postoperatively.

The quick CSF method, implemented in a 10 alternative forced-choice digit identification task, was used to assess the contrast sensitivity function34, 38. Stimuli were displayed on a gamma-corrected 46 inch LCD monitor (Model: NEC LCD P463) with a 1920×1080 pixel resolution, 50 cd/m2 mean luminance and 60 Hz vertical refresh rate. Observers viewed the display monocularly from a distance of 4 m in a dark room. For each trial, they were asked to verbally report the identities of three digits presented on the screen to the experimenter, who used the computer keyboard to enter their responses. The stimuli disappeared after all the responses were entered. Observers were given the option to report ''I don't know'' upon which the response was coded as incorrect. No feedback was provided. All three responses were used to update the posterior distribution of the CSF parameters, which in turn was used to adaptively choose the most informative combination of spatial frequency and contrast for the next trial. A new trial started 500 ms after the responses. There were 30 trials in approximately 5 min. The quick CSF data were scored to generate the cutoff spatial frequency, defined as the spatial frequency corresponding to a perceptual sensitivity of 1, and the area under the log CSF (AULCSF), a summary measure of the window to spatial vision

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the primary pterygium;
* More than 18 and less than 60 years old;
* 0.0 or better logMAR BCVA;
* The absence of other ocular disorders and no history of eye surgery and other systemic diseases.

Exclusion Criteria:

* Clinical diagnosis of recurrent pterygium or accompanied with other ocular diseases;
* less than 18 or more than 60 years old;
* The logMAR BCVA is less than 0.0;
* With the history of eye surgery and other systemic diseases.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There would have two groups included in our study, which are 40 patients of primary pterygium group and 20 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The contrast sensitivity function tested by quick CSF of the Primary Pterygium patients preoperatively | Preoperatively
  The contrast sensitivity function of the Primary Pterygium patients is lower than the normal people by qucik CSF method

SECONDARY OUTCOMES:
The contrast sensitivity function tested by quick CSF of the Primary Pterygium patients postoperatively | 1st, 3rd and 6th month postoperatively
  The contrast sensitivity function of the Primary Pterygium patients is improved compared with the normal people by quick CSF method

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yuan, Professor, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Opthalmic Center, Guangzhou, Guangdong, China